CLINICAL TRIAL: NCT01333982
Title: Evaluation of a on Community-Based Management of Neonatal Sepsis
Brief Title: Neonatal Sepsis, Evaluation, Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PR-09056
Record Dates: First submitted 2010-10-12; First posted 2011-04-12 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2011-04

CONDITIONS: Sepsis
Keywords: Neonatal Sepsis; Evaluation; Bangladesh; Drying; Wrapping; Bathing
MeSH Terms: conditions — Sepsis; Neonatal Sepsis | interventions — Amoxicillin; Gentamicins; Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Referral compliance (Experimental): Health workers will receive a basic maternal, newborn and child health training under the MNCS programme. Newborn sepsis management training will be organised for the study. The Bangladesh Perinatal Society (BPS) will take the lead in developing and implementing the training programme with support from Saving Newborn Lives (SNL) and other partners.Referral slips will be used in the intervention unions for all the sick newborns identified so that they seek care on a timely fashion.
  Interventions: Other: Amoxycillin, Gentamicin
- Neonatal sepsis (Experimental): Existing health delivery systems in the community level in managing neonatal sepsis.
  Interventions: Other: Counselling

INTERVENTIONS:
Other: Amoxycillin, Gentamicin — If referral fails, community management of neonatal sepsis according to clinical algorithm.
  Arms: Referral compliance
Other: Counselling — counselling of management of neonatal sepsis in the community according to clinical algorithm.
  Arms: Neonatal sepsis

SUMMARY:
More than half of under-five deaths in Bangladesh occur in the first month of life (neonatal period), and a substantial proportion of these deaths are due to infections (sepsis). According to the recently formulated Bangladesh National Neonatal Health Strategy (NNHS), the Government of Bangladesh is committed to improve access to quality management of neonatal infections. The strategy emphasizes that health service providers at all levels acquire the skills for managing sepsis.

Responding to the recommendations in the National Neonatal Health Strategy, this operations research seeks to evaluate alternative approaches for the management of neonatal sepsis in the community. The evaluation will focus on assessing intervention coverage, provider quality of care, and referral and referral compliance, and will undertake cost-benefit analysis of community-based neonatal sepsis management. The programme and evaluation will be within the existing health service delivery system in Bangladesh and is thus designed to inform the effective scaling up of neonatal sepsis management and contribute to the implementation of the NNHS. The interventions to be evaluated will be nested in the Maternal, Neonatal and Child Survival (MNCS) programme being implemented by the Government of Bangladesh, in partnership with and supported by UNICEF, and several national NGOs.

This operations research is being implemented by the Government of Bangladesh in collaboration with UNICEF, SNL - Save the Children (USA), Bangladesh Perinatal Society, and ICDDR,B. It will take place in four MNCS programme upazilas, where 10 unions will be randomly selected for intervention and 10 unions will be comparison. The intervention consists of training of community health workers, village doctors and health facility workers on managing neonatal sepsis in addition to essential newborn care training. In the comparison areas the health workers will only receive essential newborn care training.

The intervention and evaluation will continue for at least 18 months, with rolling surveys and two special surveys at 6 and 12 months into the project. The rolling surveys will look at intervention coverage, care-seeking, and referral and referral compliance, while the two special surveys will assess provider performance, referral compliance, and quality of care. In addition, the investigators will document implementation processes to understand what worked and what did not and why.

DETAILED DESCRIPTION:
Three to four MNCS programme upazilas will be purposively selected for this study in consultation with GoB and partners. The likely districts from where the three to four upazilas will be selected include Sunamganj, Kishoreganj, Bandarban and Sherpur. However, this may change depending on GoB/UNICEF decisions about MNCS scale-up. The upazilas will be selected considering presence of NGO partners with the ability to implement the intervention, start of MNCS in the upazilas by 2009 and no overlap with other similar programmes research projects. Twenty unions (average population of about 20,000) will be identified from the selected upazilas and randomly assigned to intervention or comparison. Unions with substantial urban populations will be excluded. In order to achieve balance in randomisation across upazilas, the investigators will make efforts to select an even number of unions from the selected upazilas.

Study design

A cluster-randomised design will be used. Of the 20 selected unions in the selected sub-districts/upazilas, 10 will be randomly assigned to intervention and 10 to comparison, that is, about 200,000 population (~40,000 households) in each arm. In both intervention and comparison unions, the common MNCS intervention package will be uniformly implemented, which includes training of community-based health workers on essential newborn care. Details of the MNCS intervention package and delivery systems can be found in Annex I. All the MNCS upazilas have also already implemented facility-based IMCI.

The objective of randomisation is to ensure balance between intervention and comparison areas in terms of population and geographical characteristics and coverage of health interventions and programmes. The sampling units (unions) will be stratified according to upazila. If any union has a total population of less then 12,000 (the minimum required to obtain an adequate sample of neonates) they will either be excluded or if such exclusion results in fewer than 20 unions being available for randomisation then two such small unions will be merged and considered as a single sampling unit. Equal number of unions for intervention or comparison will be selected from each upazila. Within each upazila, unions will be paired on distance from the upazila health complex and members of each pair be randomly selected for intervention or comparison.

In the intervention unions, in addition to routine MNCS services, services for the management of neonatal sepsis will be made available in the community, targeting all pregnant women and newborns born within the study period. Community-based management of neonatal sepsis will be provided by three types of care providers: community health workers, village doctors and community clinic care providers.

The intervention and evaluation will continue for at least 18 months. Evaluation will be ongoing and include rolling household surveys to assess intervention coverage and care-seeking and referral compliance practices. In addition, two special surveys will be conducted to assess provider performance, referral compliance, quality of care at the different levels of care, and incremental program and household costs. The first special survey will be conducted at 6 months after the implementation of the intervention and then again at 12 months. The first round of rolling survey will also include a sample of newborns born in the previous 12 months to assess baseline care-seeking patterns and coverage for neonatal sepsis.

ELIGIBILITY:
Inclusion Criteria:

* development of danger signs of neonatal sepsis during neonatal period

Exclusion Criteria:

* developing signs not in neonatal period

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20000 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Appropriate management of all cases of neonatal sepsis in the community by community level health care provider | 18 months
  Neonatal Sepsis cases, if referred, received pre-referral antibiotic and complied with referred places, or if managed on site, managed by community level health care providers trained on neonatal sepsis management and received appropriate antibiotics and minimum course of antibiotics

SECONDARY OUTCOMES:
Newborns will be dried and wrapped immediately after birth | 18 months
  Increase knowledge of caregiver regarding drying and wrapping immediately after birth
Newborns receiving breast feeding within one hour after birth | 18 months
  Increased knowledge of caregivers regarding breast feeding of newborns within one hour after birth
Newborns first bathed at least three days after birth | 18 months
  Increase knowledge of caregiver regarding first-bathing of newborns at least three days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Shams El Arifeen, MBBS, DrPh, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Sunamganj, Bandarban, Sherpur, Bāndarban, Bangladesh